CLINICAL TRIAL: NCT04803266
Title: Elective Internal Mammary Node Irradiation in Women With Node-positive Breast Cancer: a Randomized, Phase 3 Trial
Brief Title: Elective Internal Mammary Node Irradiation in Women With Node-positive Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2008-0263
Record Dates: First submitted 2021-03-09; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Internal mammary node irradiation (Experimental)
  Interventions: Radiation: Internal mammary node irradiation
- No internal mammary node irradiation (Active Comparator)
  Interventions: Radiation: No internal mammary node irradiation

INTERVENTIONS:
Radiation: Internal mammary node irradiation — Regional nodal irradiation including internal mammary node irradiation along with breast or chest wall irradiation after breast-cancer surgery
  Arms: Internal mammary node irradiation
Radiation: No internal mammary node irradiation — Regional nodal irradiation not including internal mammary node irradiation along with breast or chest wall irradiation after breast-cancer surgery
  Arms: No internal mammary node irradiation

SUMMARY:
The aim of this study is to find out whether the inclusion of internal mammary node irradiation in regional nodal irradiation improves outcomes in women with node-positive breast cancer.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized phase 3 trial. Patients with node-positive breast cancer without distant metastases were included. All patients underwent breast conservation surgery or mastectomy with axillary lymph node dissection before irradiation. Patients underwent regional nodal irradiation along with breast or chest wall irradiation and randomly allocated to either IMNI or no IMNI.

ELIGIBILITY:
Inclusion Criteria:

1. Women with histologically confirmed node-positive breast cancer who had undergone modified radical mastectomy or breast-conserving surgery and axillary dissection with ≥8 nodes removed.

Exclusion Criteria:

1. Neoadjuvant chemotherapy
2. Bilateral breast cancer
3. Distant metastasis
4. History of other malignancy
5. Involvement of supraclavicular nodes or internal mammary nodes at diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 747 (Actual)
Dates: Start 2008-11-05 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 7 years

SECONDARY OUTCOMES:
Rates of overall survival | 7 years
breast cancer-specific survival | 7 years
Number of patients with treatment-related toxicities as assessed by RTOG/EORTC Toxicity criteria and NCI CTCAE v3 | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Yong Bae Kim, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Analytic codes will be shared upon reasonable request to corresponding author.

REFERENCES:
- [Derived] Kim YB, Byun HK, Kim DY, Ahn SJ, Lee HS, Park W, Kim SS, Kim JH, Lee KC, Lee IJ, Kim WT, Shin HS, Kim K, Shin KH, Nam CM, Suh CO. Effect of Elective Internal Mammary Node Irradiation on Disease-Free Survival in Women With Node-Positive Breast Cancer: A Randomized Phase 3 Clinical Trial. JAMA Oncol. 2022 Jan 1;8(1):96-105. doi: 10.1001/jamaoncol.2021.6036. PMID 34695841